CLINICAL TRIAL: NCT01620788
Title: Randomized, Phase 3, Multicenter, Open Label, Evaluating the Effect of the Treatment of Indapamide 1.5mg/Losartan 50mg and Indapamide 1.5mg/Losartan 100mg, Compared With Hyzaar® in the Treatment of Hypertension
Brief Title: Comparison of Losartan Associated With Indapamide Versus Hyzaar® in the Hypertension Treatment
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Substancial amendment
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIEMS1111
Record Dates: First submitted 2012-05-29; First posted 2012-06-15 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Indapamide; Losartan; hydrochlorothiazide, losartan drug combination; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Indapamide 1.5mg / Losartan 50mg (Experimental)
  Interventions: Drug: Indapamide / Losartan
- Indapamide 1.5mg / Losartan 100mg (Experimental)
  Interventions: Drug: Indapamide / Losartan
- Hyzaar® (Losartan 50mg/Hydrochlorothiazide12,5mg) (Active Comparator)
  Interventions: Drug: Hyzaar®
- Hyzaar® (Losartan 100mg/Hydrochlorothiazide 25mg) (Active Comparator)
  Interventions: Drug: Hyzaar®

INTERVENTIONS:
Drug: Indapamide / Losartan — 1 tablet of Indapamide 1.5mg + Losartan 50mg, oral, a day
  Other Names: Indapamide 1.5mg / Losartan 50mg
  Arms: Indapamide 1.5mg / Losartan 50mg
Drug: Indapamide / Losartan — 1 tablet of Indapamide 1.5mg + Losartan 100mg, oral, a day
  Other Names: Indapamide 1.5mg / Losartan 100mg
  Arms: Indapamide 1.5mg / Losartan 100mg
Drug: Hyzaar® — 1 tablet of Hyzaar®, oral, a day
  Other Names: Losartan 50mg/Hydrochlorothiazide12,5mg
  Arms: Hyzaar® (Losartan 50mg/Hydrochlorothiazide12,5mg)
Drug: Hyzaar® — 1 tablet of Hyzaar®, oral, a day
  Other Names: Losartan 100mg/Hydrochlorothiazide 25mg
  Arms: Hyzaar® (Losartan 100mg/Hydrochlorothiazide 25mg)

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of indapamide 1.5mg / losartan 50mg and indapamide 1.5mg / losartan 100mg on reduction of blood pressure.

DETAILED DESCRIPTION:
* open label,randomized, multicenter
* Experiment duration: 12 weeks.
* 05 visits (day 0 - randomization), (day 1 - 2 weeks pos-randomization), (day 2 - 4 weeks pos-randomization), (day 3 - 8 weeks pos-randomization) and (day 4 - 12 weeks pos-randomization).
* evaluate the efficacy of a medication associated with two antihypertensive agents in two fixed doses compared to the Hyzaar® in patients with hypertension
* Adverse events evaluation

ELIGIBILITY:
Inclusion Criteria:

* Adults male or female aged ≥ 18 years old;
* Patients with a diagnosis of Hypertension (defined by the medical investigator) treated with monotherapy or at least two blood pressure measurements ≥ 140/90, in a sitting position with a 5' interval between measurements,
* Patients with normal lab tests results in the last six months or that the investigator consider not clinically significant,
* Patient who accept the discontinuation of previous hypertension therapy.

Exclusion Criteria:

* Patients with blood pressure ≥ 180/100 mmHg;
* Patients with uncontrolled hypertension (≥ 140/90 mmHg) treated with thiazide diuretics;
* Presence of concomitant coronary artery disease, congestive heart failure, diabetes and renal failure (creatinine> 1.5 mg / dL);
* Patients with hypo or hyperkalemia (serum potassium outside normal range);
* Patients with ALT greater than 2.5 the upper limit of normal or active liver disease;
* Pregnant women, or women in childbearing age who are not in use effective contraception or intending to become pregnant during the study period;
* Patients on drug or alcohol abuse in the last two years;
* Patients with secondary hypertension (renovascular disease, pheochromocytoma, Cushing's syndrome);
* Patients with allergic reactions or hypersensitivity to ACE inhibitors, diuretics or medications containing sulfa and / or any excipients of formulation;
* Refusal or inability to provide the Informed Consent Term.;
* Refusal to discontinue the anti-hypertensive medication.
* Patients at the discretion of the investigator does not have indication for discontinuing the current medications;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Estimated)
Dates: Start 2019-11-27 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Changes in systemic blood pressure measurements after 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Safety Will be Evaluated by the Adverse Events Occurrences | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa, Campinas, São Paulo, Brazil